CLINICAL TRIAL: NCT06340347
Title: A PHASE 1, OPEN-LABEL, SINGLE-DOSE, NON-RANDOMIZED PARALLEL GROUP STUDY TO COMPARE THE PHARMACOKINETICS, SAFETY, AND TOLERABILITY OF OSIVELOTOR (PF-07940367) IN ADULT PARTICIPANTS WITH MILD AND MODERATE HEPATIC IMPAIRMENT
Brief Title: A Study to Learn How the Body Processes the Study Medicine Called Osivelotor (PF-07940367) in People With Loss of Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C5351010; GBT601 (Other: Alias Study Number)
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Intervention Model Description: An open label, single dose, parallel cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Participants with moderate hepatic impairment will receive a single dose of osivelotor, administered orally under fasted conditions.
  Interventions: Drug: Osivelotor
- Group 2 (Experimental): Participants with mild hepatic impairment will receive a single dose of osivelotor, administered orally under fasted conditions.
  Interventions: Drug: Osivelotor

INTERVENTIONS:
Drug: Osivelotor — a single dose of osivelotor administered by mouth under fasted conditions
  Other Names:
  PF-07940367

SUMMARY:
The purpose of this study is to understand how Osivelotor is processed in people with loss of liver function.

This study is seeking participants that are:

* stable loss of liver function with mild or moderate severity
* none of underlying conditions possibly affecting the study medicine being absorbed by the body

All participants will receive one amount of Osivelotor by mouth before breakfast on the first day at the study clinic. A number of blood samples will be collected to understand how Osivelotor is changed and removed from the body. Participants will also have to undergo physical examination and other tests. This will help to understand if Osivelotor is safe.

Participants will take part in the study for a maximum of 112 days. During this time, participants will have to stay onsite for 5 days. There will be 5 study visits at the study clinic.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 16 to 40 kg/m2, inclusive; and a total body weight greater than 50 kg (greater than 110 lb)
* Stable hepatic impairment that meets the criteria for Class A or B of the Child Pugh classification with no clinically significant change in disease status within the 28 days prior to the screening visit
* Stable concomitant medications for the management of individual participants' medical history

Exclusion Criteria:

* Any condition possibly affecting drug absorption (eg, prior bariatric surgery, gastrectomy, ileal resection, prior status portacaval shunt surgery);
* Hepatic carcinoma or hepatorenal syndrome or limited predicted life expectancy;
* A diagnosis of hepatic dysfunction secondary to any acute ongoing hepatocellular process that is documented by medical history, physical examination, liver biopsy, hepatic ultrasound, computerized tomography scan, or MRI;
* Presence of clinically active Stage 3 or 4 hepatic encephalopathy. Clinically active Stage 2 encephalopathy is allowed if, in the opinion of the investigator, the participant is able to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
Area under the whole blood and plasma concentration versus time curve (AUC) from time zero (pre-dose) to the last quantifiable concentration (AUClast) of osivelotor | 0 hours (pre-dose) to 84 days post-osivelotor dose
Area under the whole blood and plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (AUCinf) of osivelotor | 0 hours (pre-dose) to 84 days post-osivelotor dose
Maximum observed whole blood and plasma concentration (Cmax) of osivelotor | 0 hours (pre-dose) to 84 days post-osivelotor dose

SECONDARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (AEs) | From baseline up to 56 days after osivelotor dose
Number of Participants With Clinically Significant Laboratory Abnormalities | From baseline up to 84 days after osivelotor dose
Number of Participants With Clinically Significant Electrocardiogram (ECG) Findings | From baseline up to 84 days after osivelotor dose
Number of Participants With Clinically Significant With Clinically Significant Vital Signs | From baseline up to 84 days after osivelotor dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Orange County Research Center, Lake Forest, California
  - Genesis Clinical Research, LLC, Tampa, Florida
  - Thomas Jefferson University-Pharmacology, Physiology and Cancer Biology, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5351010